CLINICAL TRIAL: NCT06842199
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Oral ICP-488 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy, Safety, Pharmacokinetics of ICP-488 in Patients With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-01005
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Plaque Psoriasis Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICP-488 Tablets (Experimental)
  Interventions: Drug: ICP-488 Tablets
- ICP-488 Placebo (Placebo Comparator)
  Interventions: Drug: ICP-488 Placebo

INTERVENTIONS:
Drug: ICP-488 Tablets — Eligible patients will receive ICP-488 orally as per the protocol
  Arms: ICP-488 Tablets
Drug: ICP-488 Placebo — Eligible patients will receive ICP-488 Placebo orally as per the protocol
  Arms: ICP-488 Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study to evaluate the efficacy, safety, PK characteristics of ICP-488 in Chinese adults with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following criteria:

1. Subjects voluntarily participate in this study and have signed informed consent.
2. Male or female subjects between the ages of 18 and 75 (including the threshold) at the time of signing the ICF.
3. History of plaque psoriasis ≥6 months at baseline.
4. Subjects need to receive systemic therapy and/or phototherapy.
5. The following three criteria were met: a) psoriasis Area and Severity index (PASI) score ≥12; b) Psoriasis affected body surface area (BSA) ≥10%; c) Static physician overall assessment (sPGA) ≥3 scores

Exclusion Criteria:

1. The diagnosis was non-plaque psoriasis.
2. Subjects with concurrent skin diseases that the investigator believes would interfere with the study assessments.
3. Presence of infection or immune-related disease.
4. Subjects with a history of TB or at risk for TB.
5. Received related treatment within the time window specified in the protocol.
6. An interval of less than 5 half-lives or 28 days (if any available half-life data) from the last dose of a strong CYP1A2/CYP3A4 inhibitor or inducer, or a plan to use concurrently medications with strong CYP1A2/CYP3A4 inhibitory or inductive effect during study participation.
7. The investigator has determined that there are clinically significant test results and that participation in this trial would pose an unacceptable risk to patients; Or the laboratory values of the subjects in the screening period meet the criteria specified in the protocol.
8. Pregnant or lactating women, or women who plan to become pregnant during study participation.
9. A history of severe drug allergies.
10. Any other conditions in which the investigator considers it unsuitable for the subject to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve a score of clear (0) or almost clear (1) with an improvement of at least 2 points from baseline on the static Physician's Global Assessment (sPGA) at week 16 | week 16
Percentage of subjects who achieved a PASI 75 response (a reduction of minimum 75% from baseline in PASI score) at Week 16 | Week 16

SECONDARY OUTCOMES:
Adverse events | Week 52
Percentage of subjects with PASI 50/75/90/100 in each planned visit | Week 52
Percentage of subjects with sPGA score of 0 (clear) or 1 (almost clear) and an improvement of at least 2 points from baseline in planned visits. | Week 52
The proportion of subjects with sPGA score of 0 in each planned visit. | Week 52
PK parameter: ICP-488 and its metabolite. | Week 52

CONTACTS AND LOCATIONS:
Locations (46):
- China (46):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chao-Yang Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,CMU, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Henan University of Science and technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Wuhan Hospital Of Traditional Chinese and Western Medicine (Wuhan No.1 Hospital), Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Hospital for skin diseases,Institute of dermatology chinese academy of medical sciences，peking union medical college, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Northeast International Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital skin Disease of tongji University, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School of Medicine, Jinhua, Zhejiang
  - The First Affiliated Hospital Of Ningbo University, Ningbo, Zhejiang
  - The first Affiliated hospital of Wenzhou Medical University, Wenzhou, Zhejiang